CLINICAL TRIAL: NCT02660736
Title: A Randomized, Double-blind, Single-dose, Crossover Study to Compare Two Albiglutide Drug Products for Bioequivalence in Healthy Adult Subjects
Brief Title: Bioequivalence Study of Two Albiglutide Drug Products in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201287
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Albiglutide; Randomized; Pharmacokinetics; GSK716155; Bioequivalence study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen AB (Experimental): Subjects will be receive Regimen A treatment in Session 1 followed by Regimen B treatment in Session 2.
  Regimen A: 50 mg Albiglutide Liquid Auto-injector + Placebo lyophilized DCC Pen injector.
  Regimen B: 50 mg Albiglutide lyophilized DCC Pen injector + Placebo Liquid Auto-injector.
  A minimum of an 8-week washout period between study treatment administration of Session 1 and Session 2.
  Interventions: Drug: Albiglutide Liquid Auto-injector; Drug: Albiglutide Lyophilized DCC Pen Injector; Drug: Placebo Liquid Auto-injector; Drug: Placebo Lyophilized DCC Pen injector
- Regimen BA (Experimental): Subjects will be receive Regimen B treatment in Session 1 followed by Regimen A treatment in Session 2.
  Regimen A: 50 mg Albiglutide Liquid Auto-injector + Placebo lyophilized DCC Pen injector.
  Regimen B: 50 mg Albiglutide lyophilized DCC Pen injector + Placebo Liquid Auto-injector.
  A minimum of an 8-week washout period between study treatment administration of Session 1 and Session 2.
  Interventions: Drug: Albiglutide Liquid Auto-injector; Drug: Albiglutide Lyophilized DCC Pen Injector; Drug: Placebo Liquid Auto-injector; Drug: Placebo Lyophilized DCC Pen injector

INTERVENTIONS:
Drug: Albiglutide Liquid Auto-injector — Albiglutide liquid is provided as a fixed-dose, disposable auto-injector containing albiglutide liquid (50 mg). The auto-injector delivers the study treatment in an injection volume of 1.0 mL for the 50 mg dose
Drug: Albiglutide Lyophilized DCC Pen Injector — Albiglutide is supplied as prefilled DCC Pen Injector. Each DCC contains lyophilized albiglutide 50 mg. When the injector pen product is reconstituted a neutral, isotonic solution is produced. The pen delivers albiglutide in an injection volume of 0.5 mL
Drug: Placebo Liquid Auto-injector — Liquid albiglutide matching placebo is provided as a fixed-dose, disposable autoinjector containing placebo liquid. The auto-injector delivers the placebo in an injection volume of 1.0 mL for the 50 mg placebo dose.
Drug: Placebo Lyophilized DCC Pen injector — Placebo is supplied as prefilled DCC Pen Injector. Each DCC contains matching placebo. When the injector pen product is reconstituted a neutral, isotonic placebo solution is produced. The pen delivers the placebo in an injection volume of 0.5 mL.

SUMMARY:
Albiglutide (Alb) is a novel analogue of glucagon-like peptide-1 (GLP-1) has been developed and approved for the treatment of type 2 diabetes mellitus. Currently, lyophilized albiglutide and the diluent are provided in a dual chamber Cartridge (DCC) single-dose pen injector, requiring reconstitution prior to use. A liquid formulation of albiglutide will enable the use of a liquid product in a ready-to-use single dose auto-injector. To support the development of the liquid auto-injector product, this healthy volunteer bioequivalence study will be conducted to compare the liquid drug product to the currently available lyophilized product. This is Phase I, randomized, double-blind, double dummy, single-dose, 2-period crossover study in healthy volunteers. This study will compare the pharmacokinetics and safety of the albiglutide 50 mg liquid drug product with the albiglutide 50 mg commercial lyophilized drug product.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age.
* Healthy.
* Subject is a nonsmoker.
* Subject's body mass index (BMI) is >=18 kilogram/meter square (kg/m^2) and <=30 kg/m^2
* Male or
* Female

Exclusion Criteria:

* Alanine aminotransferase (ALT) >1.5 x upper limit of normal range (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 millisecond (msec).
* Systolic blood pressure is >=140 millimeter of mercury (mmHg) at Screening;
* Diastolic blood pressure is >=90 mmHg at Screening;
* Heart rate is >100 beats/min at Screening.
* estimated glomerular filtration rate (eGFR) <=80 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) at Screening.
* Fasting triglyceride level >300 milligram per deciliter (mg/dL) at Screening.
* History of significant cardiovascular or pulmonary dysfunction prior to Screening.
* History of thyroid dysfunction or an abnormal (i.e., outside the normal reference range) thyroid function test assessed by thyroid stimulating hormone at Screening.
* History of gastrointestinal surgery that could influence gastric emptying (e.g., gastrectomy, gastric bypass).
* History of pancreatitis.
* Personal or family history of multiple endocrine neoplasia type 2.
* Personal or family history of medullary carcinoma of the thyroid.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days.
* History of regular alcohol consumption within 6 months of the study.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* Subject has previously received any GLP-1 mimetic compound (eg., exenatide, liraglutide, lixisenatide, dulaglutide).
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Subject has donated blood in excess of 500 mL within 56 days prior to dosing or intention of donating in the month after completing the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from 0 to the last measurable concentration (AUC 0-t) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide plasma concentrations and (AUC 0-t).
AUC from 0 to infinity (AUC [0-inf]) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide plasma concentrations AUC(0-inf).
Peak plasma concentration (Cmax) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide Cmax.

SECONDARY OUTCOMES:
Time to maximal concentration (Tmax) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide Tmax.
Clearance (CL/F) for albiglutide in session 1 and 2. | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide CL/F
Volume of distribution (V/F) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2
  PK blood samples will be collected for determination of albiglutide V/F
Number of subjects with adverse events (AE) and clinical observations as a measure of safety and tolerability | Up to 21 weeks
  AE will be collected during the study. Intensity of AE will be captured
Safety as assessed by 12-lead electrocardiogram (ECG) | Screening, Day -1, Day 4, and Day 35 in both sessions 1 and 2
  Single 12-lead ECGs will be obtained at the specified time points during the study using an ECG machine that automatically calculates the heart rate and other measures.
Safety as assessed by systolic, diastolic blood pressure, and pulse rate measurements | Up to 21 weeks
  Systolic and diastolic pressure and pulse rate will be measured at specified time point
Immunogenicity as assessed by enzyme-linked immunosorbent assay (ELISA) and hypersensitivity reactions. | Day 1 in both sessions and Day 13 in session 1 and follow-up visit
  Immunogenicity serum samples will be collected at specified time points to assess the presence of anti-drug antibodies through enzyme-linked immunosorbent assay (ELISA) method.
Half-life (T1/2) for albiglutide in session 1 and 2 | Predose (0), 24, 48, 72, 96, 120, 216, 312, 480, 672, and 840 hours post-dose in both sessions 1 and 2.
  PK blood samples will be collected for determination of albiglutide T1/2.
Composite of hematology parameters as a measure of safety | Up to 21 weeks
  The following hematology parameters will be measured: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, Reticulocyte count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), MCH Concentration, white blood cell (WBC) count, neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Composite of clinical chemistry parameters as a measure of safety | Up to 21 weeks
  The following clinical chemistry parameters will be measured: blood urea nitrogen (BUN), creatinine, fasting glucose, uric acid, thyroid-stimulating hormone (TSH), potassium, sodium, calcium, phosphorus, magnesium, aspartate amino transferase (AST), alanine amino transferase (ALT), alkaline phosphatase, gamma glutamyl transferase (GGT), chloride, total and direct bilirubin, total protein, albumin, total carbon dioxide, and fasting triglycerides.
Composite of urinalysis parameters as a measure of safety | Up to 21 Weeks
  The following urinalysis parameters will be measured: specific gravity, power of hydrogen (pH), glucose, protein, blood and ketones by dipstick; microscopic examination (if blood or protein is abnormal), microalbumin, creatinine, albumin/creatinine ratio, blood, leukocyte esterase, and nitrites.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Derived] Shaddinger BC, Vlasakakis G, Soffer J, Thorpe KM, Hatch D, Nino AJ. A Randomized, Double-Blind, Single-Dose, Crossover Study to Demonstrate the Bioequivalence of 2 Formulations of Albiglutide in Healthy Adult Participants. Clin Pharmacol Drug Dev. 2019 Apr;8(3):361-370. doi: 10.1002/cpdd.606. Epub 2018 Jul 31. PMID 30063297